CLINICAL TRIAL: NCT06979726
Title: Gator SCALES-WHF: SubCutaneous Administration of Lasix to Eliminate Symptoms of Worsening Heart Failure
Acronym: GatorScalesWHF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: SQ Innovation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202500547
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure; Volume Overload
MeSH Terms: conditions — Heart Failure; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lasix ONYU (Other): Patients receiving Lasix ONYU
  Interventions: Drug: Lasix ONYU

INTERVENTIONS:
Drug: Lasix ONYU — Providing subcutaneous furosemide to eligible patients

SUMMARY:
The primary objective of the study is to develop, implement, and evaluate a site-specific clinical pathway for at-home treatment of eligible patients presenting to the clinic with worsening heart failure.

The secondary objectives are:

1. To evaluate patient factors related to parenteral decongestion at home.
2. To evaluate the safety and device operation of Lasix ONYU treatment under circumstances that mimic real-world use.
3. To identify opportunities for process improvement before the routine implementation of the new clinical pathway.

DETAILED DESCRIPTION:
The investigators will conduct an open-label, non-comparative, real-world study to evaluate the effectiveness and feasibility of at-home decongestion treatment using Lasix ONYU in patients with worsening heart failure (WHF). During a clinical visit at the UF Heart Failure Clinic, Emergency Department, or Clinical Decision Unit, the study assess whether a patient meets eligibility criteria for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above
2. Previously diagnosed with Congestive Heart Failure (HFpEF or HFrEF)
3. Fluid overload due to worsening HF requiring parenteral diuretic treatment as assessed by at least 2 of the following:

   1. BNP > 200
   2. JVP > 10cmH20
   3. Presence of S3
   4. LE Edema
   5. Weight gain of > 5lbs in the past 5 days
4. Failed oral uptitration of loop diuretic over the prior 5 days or presented with symptoms too advance to justify additional oral uptitration attempts to resolve congestion symptoms.
5. Expected to require a minimum of three days of parenteral diuretic treatment
6. Written informed consent
7. Able and willing to operate Lasix ONYU and comply with study requirements or has a caregiver who can assume these roles.

Exclusion Criteria:

1. Age above 80 years
2. Unable or unwilling to provide informed consent.
3. Any medical condition or circumstances that would require further clinical investigation or hospitalization
4. Presence or history of electrolyte abnormalities that may be exacerbated by parenteral loop diuretic treatment
5. Home or current living environment not suitable for outpatient management and diuresis
6. Pregnant or breastfeeding
7. Unable to comply with clinic-required follow up procedure
8. Baseline chronic renal disease with CKD Stage V
9. Any surgical or medical condition which, in the opinion of the investigator, may pose an undue risk to the subject, interfere with participation in the study or which may affect the integrity of the data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Lasix ONYU Use | 30 days
  Adverse reactions, acute kidney injury

SECONDARY OUTCOMES:
Hospital Readmission | 30 days
  30 day readmission from time of Lasix ONYU administration

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States